CLINICAL TRIAL: NCT02320825
Title: Phase III Multicenter Randomized Study Comparing Local Tumor Control After Post-Operative Single-Fraction or Hypofractionated Stereotactic Radiosurgery in the Treatment of Spinal Metastases
Brief Title: Randomized Study Comparing Local Tumor Control After Post-Operative Single-Fraction or Hypofractionated Stereotactic Radiosurgery in the Treatment of Spinal Metastases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Johns Hopkins University (Other); Massachusetts General Hospital (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-233
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-01

CONDITIONS: Spinal Metastases
Keywords: Stereotactic Radiosurgery (SRS); Single-Fraction; Hypofractionated; Spinal surgery; 14-233

ARMS (2):
- single-fraction SRS (24 Gy) (Experimental): single-fraction (24Gy) SRS within eight weeks of having undergone spinal decompression surgery.
  Interventions: Radiation: single-fraction SRS; Behavioral: Quality of Life Measures
- high-dose hypofractionated SRS (27 Gy in 3 fractions) (Experimental): hypofractionated (3 fractions of 9Gy, total dose of 27Gy) SRS within eight weeks of having undergone spinal decompression surgery.
  Interventions: Radiation: high-dose hypofractionated SRS; Behavioral: Quality of Life Measures

INTERVENTIONS:
Radiation: single-fraction SRS
  Arms: single-fraction SRS (24 Gy)
Radiation: high-dose hypofractionated SRS
  Arms: high-dose hypofractionated SRS (27 Gy in 3 fractions)
Behavioral: Quality of Life Measures

SUMMARY:
The purpose of this study is to find out whether giving one higher dose of radiation is as good at treating the tumor in the patient's spine after surgery as giving three lower doses of radiation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed metastatic cancer (Diagnosis made or confirmed at MSKCC for MSKCC participants. Institutional pathologic determination accepted from participating multicenter sites.)
* Age ≥18 years
* Life expectancy ≥3 months
* ECOG ≤ 3
* Spinal surgery carried out with the goal of spinal cord decompression and spinal stabilization within 8 weeks
* Post-operative CT myelogram or MRI perfusion with evidence of separation of tumor and the spinal cord It should be noted that patients with multiple lesions will be eligible as long as there are no overlapping fields of radiation, including at various time frames.

Exclusion Criteria:

* Primary spine tumor
* Age < 18
* Pregnancy
* Lack of adequate (≥ 2 mm) separation between the spinal cord and the tumor on post-operative CT myelogram or MRI perfusion
* Radiosensitizing chemotherapy (taxol, taxotere, cisplatin, gemcitabine, 5-fluorouracil) given within one week of radiation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12-16 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Laufer, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Stanford University Medical Center, Stanford, California
  - John Hopkins Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- High-dose Hypofractionated SRS (27 Gy in 3 Fractions): hypofractionated (3 fractions of 9Gy, total dose of 27Gy) SRS within eight weeks of having undergone spinal decompression surgery.
  high-dose hypofractionated SRS
  Quality of Life Measures
- Single-fraction SRS (24 Gy): single-fraction (24Gy) SRS within eight weeks of having undergone spinal decompression surgery.
  single-fraction SRS
  Quality of Life Measures
Period: Overall Study
Arm/Group | High-dose Hypofractionated SRS (27 Gy in 3 Fractions) | Single-fraction SRS (24 Gy)
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-dose Hypofractionated SRS (27 Gy in 3 Fractions) | Single-fraction SRS (24 Gy) | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Full Range); unit: years] | 55.125 [45 to 72] | 59.75 [46 to 71] | 57.44 [45 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 7 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Local Tumor Control Using MRI or CT
Description: will be radiographically determined according to routine standard of care post-surgical and post-treatment imaging (MRI or CT) of the spine. Local tumor control will be defined as the lack of local tumor progression at the irradiated site on follow-up imaging.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Single-fraction SRS (24 Gy) | High-dose Hypofractionated SRS (27 Gy in 3 Fractions)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Treatment-related Toxicity Using CTCAE v4.0
Description: Adverse events will be assessed by the investigators according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Single-fraction SRS (24 Gy) | High-dose Hypofractionated SRS (27 Gy in 3 Fractions)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Quality of Life Between the Two Cohorts Determined Through Patient-reported Responses of the BPI
Description: will be determined through patient-reported responses of the BPI. Pain severity at its worst (question #5) and the average of the pain interference (average of question #9)
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Single-fraction SRS (24 Gy) | High-dose Hypofractionated SRS (27 Gy in 3 Fractions)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | High-dose Hypofractionated SRS (27 Gy in 3 Fractions) | Single-fraction SRS (24 Gy)
All-Cause Mortality (participants affected / at risk) | 7/8 | 5/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-dose Hypofractionated SRS (27 Gy in 3 Fractions) (N=8) | Single-fraction SRS (24 Gy) (N=8)
Esophagitis (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT02320825/Prot_SAP_000.pdf